CLINICAL TRIAL: NCT04957589
Title: The Effect of a Very Low Calorie Diet (VLCD) With and Without Concomitant High Intensity Interval Training (HIIT) on Muscle Protein Synthesis (MPS) in Middle-aged Overweight Diabetic Men
Brief Title: VLCD & Adjuvant Exercise Effect in Overweight Diabetic Men
Acronym: VLCDeXDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19026_CMMP; 255016 (Other: IRAS)
Record Dates: First submitted 2020-06-05; First posted 2021-07-12 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus Type 2 in Obese
MeSH Terms: interventions — Caloric Restriction; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This is a proof-of-concept, single centre, randomised, non-blinded control trial.
Masking Description: Masking is infeasible, as the participants will know which intervention they are partaking in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLCD & HIIT (Experimental): Very low calorie diet (standardised LighterLife meal replacement packages consisting of approximately 150kcal each, amounting to 600kcal/day, with 200kcal of a pre-determined free expenditure consisting of nuts and/or vegetables) High intensity interval training (3x sessions per week following intensity estimation using cardiorespiratory testing (VO2max), using an established training protocol within our department) No additional protein supplementation
  Interventions: Dietary Supplement: Very Low Calorie Diet; Other: High Intensity Interval Training
- VLCD only (Active Comparator): Very low calorie diet (standardised LighterLife meal replacement packages consisting of approximately 150kcal each, amounting to 600kcal/day, with 200kcal of a pre-determined free expenditure consisting of nuts and/or vegetables) No additional exercise or protein supplementation
  Interventions: Dietary Supplement: Very Low Calorie Diet

INTERVENTIONS:
Dietary Supplement: Very Low Calorie Diet — A dietary intervention consisting of four meals (provided by LighterLife®), totaling approximately 600kcal/day (each meal comprising approximately 150kcal/day). Participants are provided with a choice of one of six "meal protocols", which consist of a pre-set combination of meals that arrive at approximately 52g protein, more than 15g fibre and less than 20g sugar per day.
  Other Names: LighterLife®; Very Low Energy Diet; Calorie Restriction; Caloric Restriction
Other: High Intensity Interval Training — The HIIT training will consist of a five-exercise approach across three movements (star jumps, standing squats, on-the-spot-sprinting, standing squats and star jumps), which are collectively described as a cycle in this context. Each exercise is performed for 60 seconds with a 90 seconds recovery period. Each training session will begin with a two minute warm-up and cooldown (on-the-spot-jogging) followed by five minutes of static stretching. Volunteers would aim to exceed the initial number of star jumps and standing squats in the subsequent attempt per cycle. A total of three training sessions per week are to be completed, preferably non-consecutive but may be consecutive on no more than two training sessions per week. Progression is through a gradual increase in volume (repetitions of star jumps and standing squats) on a per-session basis.
  Other Names: HIIT; Home HIIT
  Arms: VLCD & HIIT

SUMMARY:
Sarcopenia is defined as the incremental age-related loss of skeletal muscle in humans which generally begins from forty years old. It is associated with an overall reduction in quality of life and increased morbidity and mortality. Patients with type two diabetes mellitus (T2DM) are particularly at risk of developing sarcopenia, partly due to the condition and also due to the common incidence after or during middle age. A promising recently-investigated and effective conservative approach to T2DM is through very low calorie diets (VLCD). Some studies have shown that the diabetic status of some patients can be reversed through VLCD. However, VLCD will theoretically result in an acceleration of sarcopenia. This presents as a limiting factor for the implementation of VLCD in this at-risk patient group. Skeletal muscle tissue is encouraged to grow in size or be maintained through two means - an increase in circulating protein breakdown products, or through resistance exercise (RE). Additionally, RE has been shown to increase the body's sensitivity to insulin, the main hormone which controls circulating glucose levels and is frequently impaired in T2DM, as well as temporarily decreasing glucose levels. The precise mechanism by which these happen is not fully understood yet. In this study, the effect of a VLCD is used, alongside one form of exercise (high intensity interval training, HIT), in overweight, middle-aged male patients with T2DM. 10 patients are to be recruited into each group (control/VLCD-only and VLCD with HIT) at our centre. Patient weight, markers of muscle protein synthesis, glucose levels and changes to blood vessels will be investigated before, during and after across a six week timeframe. Investigations will include muscle and fat biopsies, blood samples, ultrasound scans, strength testing and deuterium oxide (D2O) isotope ingestion for later non-invasive body fluid sample mass spectrometric analysis.

DETAILED DESCRIPTION:
Very low calorie diet (VLCD) is increasingly being utilized to improve cardio-metabolic outcomes in overweight/obese individuals with type 2 diabetes mellitus (T2DM), but concerns regarding its association with skeletal muscle mass losses persist, especially in middle-aged/older individuals, who are already at risk of accelerated sarcopenia. This is particularly relevant in people at risk of developing diabetes due to the rising incidence and prevalence of diabetes among older patients as well as accelerated sarcopenia in diabetes compared with non-diabetes. Given that low skeletal muscle mass and function is linked to mortality, frailty, and adverse cardio-metabolic outcomes, increased understanding of the mechanisms of VLCD-induced muscle atrophy, and novel strategies to overcome this is crucial to optimize healthy ageing. Alongside nutrition, physical activity is another key driver of muscle protein synthesis, with habitual physical activity required to maintain muscle mass. A number of studies have shown that even short-term muscle disuse (or reduced use in the form of reduced ambulation (e.g. 2 weeks of <1500 steps/day) or limb immobilization causes muscle wasting. Exercise has also been shown to improve metabolic control by increasing muscle glucose uptake during muscle contractions via insulin-independent mechanisms, and also by increasing skeletal muscle insulin sensitivity following physical activity. HIT has been shown in a number of studies to improve both cardiovascular and metabolic function in a variety of cohorts. Therefore, this study aims to quantitatively determine whether HIT helps prevent a major physiological detrimental effect of VLCD.

This study will randomise volunteers to:

1. VLCD ("Lighter Life" meal replacement product, total 600 calories (kcal)) alone (200kcal free allowance) (N=10)
2. VLCD and HIT (200kcal free allowance) (N=10) This will be undertaken in overweight and obese patients (BMI=27-50kg/m2) of male gender and between the ages of 35-65 years. Based on a power calculation derived from recently-published trial data utilising VLCDs and with MPS as the primary outcome, a minimum of 8 participants per group would be sufficient, with a further N=2 per arm (an increase in 25%) implemented to account for drop-outs.

The study will aim to recruit (to allow for potential non-completion) 10 subjects per group. Volunteers would undergo detailed physiological and metabolic investigations before and after interventions

1. Skeletal muscle mass, function and protein metabolism
2. Vascular function (microvascular perfusion, macrovascular blood flow and endothelial function)
3. Cardio-metabolic status (glucose handling, cardiorespiratory function, central blood flow parameters)
4. mechanisms regulating changes in glucose handling and muscle protein turnover It is anticipated that HIT may ameliorate VLCD-induced reductions in skeletal muscle mass and function, by boosting the molecular signals which involve the retention of muscle mass. This adjuvant exercise interventions may also elicit improvements in cardio-metabolic health (vs. VLCD alone) via improvements in blood vessel function.

The findings from this project could enhance our understanding on the role of VLCD in inducing improvement in cardio-metabolic health, provide rapid, practical low cost clinical interventions for people with T2DM and/or obesity, while unearthing potential new therapeutic targets for the future management of high blood sugar and obesity in people with T2DM.

STUDY PROTOCOL After having passed screening and being formally enrolled, participants will be randomised and stratified (described previously), and then attend the department twice prior to their intervention commencement, with each day consisting of a full study day, whereby the various primary and secondary outcome measurements will be performed.

On the first study day (D-5 from intervention), subjects will be asked to fast from midnight (except for water). This first 'study day' will consist of, in chronological order, repeat height and weight measurement, a baseline urine sample, DXA and oral glucose tolerance test (OGTT) with concurrent questionnaire completion, followed by lunch. This is followed by hand grip dynamometry, electromyogram, maximal voluntary isometric contraction (MVC), the Short Physical Performance Battery (SPPB), and 1 repetition-maximum (1RM) testing of three lower body (leg press, hamstring curl, quadriceps extension) and three upper body movements (chest press, machine row, machine pulldown). Thereafter, participants would be fitted with an Actiheart monitor, followed by a staggered dosing of a D2O bolus with a concurrent bolus dose of D3-creatine. Additionally, they would be provided with several collection vessels (24 hour jar, two collection pots for 48 hour and 72 hour spot samples for the D3-creatine; a saliva collection pot to be filled two hours following the D2O bolus). They would also be provided with a loading dose of 3-methylhistidine (3MH) to be taken one day prior to the second study day (D-1 from intervention). Finally, they would be provided with an updated itinerary of the available VLCD meals for selection.

Between the two study days (D-4 to D-1 from intervention), the participant would collect their D3-creatine-containing urine at home (24 hour period, and 48 & 72 hour spot samples). Additionally, one day prior to the second study day (D-1 from intervention), participants would be asked to consume the 3MH bolus at precisely 13:00. During the interim period, the participant would also be contacted to receive their preferences for meal profiles, which would be organised by the department. Finally, if the participant had been randomised into the 'VLCD only' group, they will advise the research team of their preferred food items (vegetables and/or nuts) during this interval, in order for a calculation of the approximate breakdown of calories that may be required to achieve a 200kcal value.

On the second study day (D0 from intervention), subjects would once again be asked to fast from midnight (except for water). Upon attendance, they would be asked to provide a fasting saliva sample, blood (a repeat of the screening panel, alongside the '0 hour' serum 3MH level and D2O baseline measurement). Additionally, they would have their estimated 50% 1RM calculated for the quadriceps leg extension of their dominant leg (for utilisation in the subsequent analyses that day). They will also be expected to return their Actiheart monitor and D3-creatine samples for subsequent analysis.

Thereafter, the participants would undergo (in chronological order) abdominal adipose tissue biopsy, vastus lateralis muscle biopsy (non-dominant leg), vastus lateralis ultrasound assessment (dominant leg), contrast-enhanced ultrasound scan (using the Sonovue agent; dominant leg), leg blood flow (dominant leg), flow-mediated dilation (dominant arm), and cardiopulmonary exercise testing (CPET). Throughout, across a four hour period from 09:00 to 13:00, serial measurement of the participant's serum 3MH levels are performed. At the end of the session, the participant would be provided with two to three weeks of VLCD meals (per their previously-agreed profile choices pending availability), alongside a diet and sleep diary. Further, they will be provided with the details of a registered dietician for support, and six once-weekly 'top up' doses of D2O, with the adjoining saliva sample vessels, to be filled immediately prior to 'top up' and two hours afterwards.

The day after, the participant will commence their VLCD diet (D1), and will be expected to attend the department for a brief period several days afterwards (D4-5) for an inspection of their biopsy incision sites by a research clinician.

Within weeks three to four of the intervention, a peri-intervention study day will be undertaken, whereby the participant would have repeat serial 3MH testing (as described in the second pre-intervention study day), alongside another set of repeat blood tests (as described in the first pre-intervention study day). All D2O saliva samples generated up to this juncture may be submitted to us at this time. The participant would also be refitted with an Actiheart monitor, to be worn for five full days.

Following the completion of six full weeks of interventionIn the sixth and final week of their intervention period, the participants would be brought in for the post-intervention study days, which fully replicate the procedures described in the pre-intervention study days, with the exception of a D2O loading dose, and the returning of the Actiheart monitor worn following the peri-intervention study day. Thus, these final two post-intervention study days would occur on week six day two and week six day seven of the intervention period.

After the post-intervention study days have been completed, the participant would once again attend the department after several days for a biopsy site incision inspection, in addition to the organisation of their reimbursement and guidance with respect to transitioning towards an increased calorie intake post-intervention All subjects will have 6-week intervention period of VLCD nutritional intervention with LighterLife VLCD meal replacement diets, 600kcal/day with 100% recommended daily allowance (RDA) vitamins and minerals. Meal replacements, which will be acquired from LighterLife, comprise of four food packs a day in the forms of soups, porridge, bars and drink mixes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide informed consent.
* Adult patients between the age of 30-65 years
* A body mass index (BMI) of between 27-50
* Confirmed Type 2 Diabetes Mellitus (T2DM)

Exclusion Criteria:

* contrast (Sonovue) sensitivity,
* known renal, musculoskeletal, neurological, bowel, cardiovascular, respiratory or cerebrovascular disease,
* or current/recent formal exercise regime participation (within two years).
* Prospective volunteers with a weight exceeding 120kg are ineligible to participate due to the weight restriction present in the DEXA machine.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis (MPS) | 6 weeks (throughout intervention)
  Estimation via weekly sampling of saliva following deuterium oxide (D2O) tracer solution administration relative to baseline.
Muscle Protein Breakdown (MPB) (3MH) | 6 weeks (one day prior to intervention study dates in pre, peri and post periods)
  Estimation via peri-intervention study date measurement of serum and urine 3-methylhistidine (3MH) concentration relative to baseline.

SECONDARY OUTCOMES:
Vascular function (femoral artery blood flow) | 6 weeks (pre and post intervention study dates only)
  Macrovascular assessment of femoral artery blood flow, assessed pre- and post- leg extension in the participant's dominant leg.
Vascular function (contrast enhanced ultrasound scan) | 6 weeks (pre and post intervention study dates only)
  Microvascular assessment of the vastus lateralis muscle in the participant's non-dominant leg using ultrasound scanning and Sonovue contrast agent.
Vascular function (brachial artery reactive hyperaemia) | 6 weeks (pre and post intervention study dates only)
  Microvascular assessment of the brachial artery's endothelial response to transient ischaemia through the application of a fixed cuff and an assessment of the wave-forms.
Body composition (Dual-Energy X-ray Absorptiometry (DEXA) scan) | 6 weeks (pre and post intervention study dates only)
  Assessment of participant body composition, including total mass, fat mass, lean body mass, and adipose tissue deposition pattern changes.
Body composition (body weight measurement) | 6 weeks (pre and post intervention study dates only)
  Measurement of participant weight (in kg).
Body composition (body mass index (BMI) estimation) | 6 weeks (pre and post intervention study dates only)
  Calculation of participant BMI using Outcome 7 and the participant's height from screening.
Muscle structure (vastus lateralis cross-sectional area) | 6 weeks (pre and post intervention study dates only)
  Measured through external ultrasound scanning.
Muscle structure (vastus lateralis pennation angle) | 6 weeks (pre and post intervention study dates only)
  Measured through external ultrasound scanning.
Muscle structure (vastus lateralis circumference) | 6 weeks (pre and post intervention study dates only)
  Measured through external ultrasound scanning.
Muscle structure (vastus lateralis fascicle length) | 6 weeks (pre and post intervention study dates only)
  Measured through external ultrasound scanning.
Muscle function (1-repetition maximum assessment) | 6 weeks (pre and post intervention study dates only)
  1-repetition maximum strength assessment in the bench press, cable row, lat pulldown, leg press, leg curl, leg extension: performed through several supervised warming-up exercise sets each, followed by a single maximum effort set, with the 1-repetition maximum calculated thereafter.
Muscle function (maximum voluntary contraction) | 6 weeks (pre and post intervention study dates only)
  Assessment of voluntary contraction of the quadriceps muscle.
Metabolic status (Oral glucose tolerance testing (OGTT)) | 6 weeks (pre and post intervention study dates only)
  Undertaken to assess for insulin sensitivity and resistance.
Metabolic status (screening blood testing via venepuncture) | 6 weeks (pre and post intervention study dates only)
  Repeat of screening blood battery testing (full blood count, urea and electrolytes, liver function test, thyroid function test, lipid profile). In each instance, the results are compared against the local laboratory reference range for the respective physiological parameters.
Metabolic status (mitochondrial respiration) | 6 weeks (pre and post intervention study dates only)
  Assessed via sampling of muscle tissue (vastus lateralis) via biopsy. Sample processed using Oroboros Instruments O2k machine. Oxygen consumption rate calculated.
Cardiopulmonary fitness | 6 weeks (pre and post intervention study dates only)
  Ergometer-based assessment of VO2max
Skeletal Muscle & Creatine Pool Assessment (D3-C) | 6 weeks (pre and post intervention study dates only)
  Total-body creatine pool size and skeletal muscle mass determination using D3-Creatine (D3-C).

CONTACTS AND LOCATIONS:
Overall Officials: Iskandar Idris, BMBS FRCP DM, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant medical information obtained as a result of this study are considered confidential and disclosure to third parties is prohibited with the exceptions noted above.
  Such medical information may be given to the participant's medical team and all appropriate medical personnel responsible for the participant's welfare.
  If information is disclosed during the study that could pose a risk of harm to the participant or others, the researcher will discuss this with the Chief Investigator (CI) and where appropriate report accordingly.
  Data generated as a result of this trial will be available for inspection on request by the participating physicians, the University of Nottingham representatives, the local Research Ethics Committee (REC) and the regulatory authorities.
  Elements of the results from this study will be submitted for peer-review in at least one publication.